CLINICAL TRIAL: NCT06874348
Title: Functional MRI During Resting State in Patients with Eating Disorders: a Longitudinal Prospective Study on Neuropsychopathological Correlates
Brief Title: Functional MRI During Resting State in Patients with Eating Disorders
Status: Recruiting | Type: Observational
Sponsor: Meyer Children's Hospital IRCCS (Other)
Collaborators: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Sponsor
Other Study IDs: RS-FMRI-ED
Record Dates: First submitted 2025-02-27; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Anorexia Nervosa; Bulimia Nervosa
Keywords: resting state fMRI; longitudinal evaluation
MeSH Terms: conditions — Anorexia Nervosa; Bulimia Nervosa | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Anorexia Nervosa - minors
  Interventions: Diagnostic Test: structural and functional MRI
- Bulimia Nervosa - minors
  Interventions: Diagnostic Test: structural and functional MRI
- Anorexia Nervosa - adults
  Interventions: Diagnostic Test: structural and functional MRI
- Bulimia Nervosa - adults
  Interventions: Diagnostic Test: structural and functional MRI

INTERVENTIONS:
Diagnostic Test: structural and functional MRI — structural and functional MRI

SUMMARY:
The goal of this observational study is to learn if clinical and neurophysiological characteristics dynamics may follow similar trends in a longitudinal characterization of patients with a diagnosis of an eating disorder.

The primary hypothesis is that the reversal of Functional Magnetic Resonance Imaging (fMRI) baseline alternations is positively associated with symptomatic amelioration.

The secondary hypothesis is that the degree of (f)MRI baseline alternations is positively associated with symptoms.

Participants will be asked to complete psychometric questionnaires, perform a fMRI and be recalled at 12 months for a follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Age between 12 and 40 years old
* Current diagnosis of Anorexia Nervosa or Bulimia Nervosa according to DSM-5-TR.

Exclusion Criteria:

* Previous or current diagnosis of schizophrenia or bipolar disorder,
* Acute psychosis
* Substance abuse
* Severe medical comorbidities (hypercapnia, severe hypertension, cardiac arrhythmia, organ failure)
* incapacity to grant written or verbal consent

Ages: 12 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Anorexia Nervosa or Bulimia Nervosa patients between 12 and 40 years old
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in cortical thickness | baseline, 12 months post-enrollment
Weight restoration | baseline - 12 months post-enrollment
Child Behavior Checklist (CBCL) score | Baseline - 12 months post enrollment
Children's Depression Inventory (CDI) score | baseline, 12 months post-enrollment
Multidimensional Anxiety Scale for Children (MASC) | Baseline - 12 months post-enrollment
Eating Disorder Inventory (EDI) psychometric score | Baseline - 12 months post-enrollment

SECONDARY OUTCOMES:
Change of measure of interhemispheric connectivity between corresponding areas in fMRI (Voxelwise Homotopic Connectivity - VMHC) | baseline, 12 months post-enrollment
  VMHC is a measure of interhemispheric connectivity between corresponding areas in fMRI. VMHC measures the level of symmetry, or correlation, between left/right pairs of voxels or brain areas.
Change in Regional Homogeneity (ReHo) index | baseline, 12 months post-enrollment
Chiange in amplitude of low-frequency fluctuations (ALFF) and fractional amplitude of low-frequency fluctuations (fALFF) of the blood oxygen-level dependent (BOLD) signal in fMRI data | baseline, 12 months post-enrollment
Change in connection degree between each node and other nodes (Degree of Centrality - DC) in the network in the brain. | Baseline - 12 months post-enrollment

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Azienda Ospedaliero-Universitaria Careggi, Firenze, Florence
  - Meyer Children's Hospital IRCCS, Florence

IPD SHARING:
Plan to Share IPD: No